CLINICAL TRIAL: NCT05289336
Title: DAHANCA 27 Transoral Laser Microsurgery for T1a Glottic Cancer
Acronym: DAHANCA 27
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danish Head and Neck Cancer Group (Network)
Responsible Party: Principal Investigator, Jens Overgaard, Professor, MD, Danish Head and Neck Cancer Group
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DAHANCA 27
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Glottic T1
Keywords: Transoral laser microsurgery; Accelerated radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Phase 2 prospective non-inferiority trial comparing with previous prospective collected national cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transoral Laser Microsurgery (Experimental): Transoral Laser Microsurgery
  Interventions: Procedure: Transoral Laser Microsurgery

INTERVENTIONS:
Procedure: Transoral Laser Microsurgery

SUMMARY:
To evaluate whether Transoral Laser Microsurgery (TLM) is non-inferior compared to Accelerated Radiotherapy (accRT) in the treatment of T1aN0M0 glottic SCC

DETAILED DESCRIPTION:
Since 2003 the Danish national standard treatment for T1aN0M0 glottic SCC has been accelerated RT (66Gy. 2 GY/fraction, 6 fractions/week). In 2012 cordectomy type I-III using TLM was introduced as an experimental treatment.

The DAHANCA 27 trial is a comparative non-inferiority phase II study comparing two timely separated national patient cohorts. Patients treated with radical TLM from September 2012 to April 2016 were included in the TLM cohort, and patients treated with accelerated RT from January 2003 to august 2012 were included in the RT cohort

ELIGIBILITY:
Inclusion Criteria:

* Danish patients aged ≥18 years diagnosed with a T1aN0M0 glottic squamous cell carcinoma (SCC)

Exclusion Criteria:

* Unable to complete curative intended protocol treatment and/or planned follow up
* informed concent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
laryncegtomy free survival | 5 years
  Alive with larynx

SECONDARY OUTCOMES:
Local control | 5 years
  Free from disease after primary treatment
Ultimate tumor control | 5 years
  Free from disease after primary treatment including salvage RT or surgery
Overall survival | 5 years
  Death of any cause
Voice quality | 3 years
  Voice Handicap Index score
Radiation free survival | 5 years
  survival without being treated with RT
any other treatment related morbidity | 5 years
  Dahanca morbidity recording

CONTACTS AND LOCATIONS:
Overall Officials: Nina M Lyhne, MD, Study Chair — Aalborg University Hospital, Denmark
Locations (5):
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Department of Experimental Clinical Oncology, Aarhus University Hospital, Aarhus
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided
information can be obtained from the Dahanca database, pending legal and dataprotection accept and relevance